CLINICAL TRIAL: NCT05576324
Title: Effect of the CFTR-modulating Triple Therapy Elexacaftor - Tezacaftor - Ivacaftor on Numerical Distribution in Peripheral Mononuclear Immune Cells Derived From Patients With Cystic Fibrosis
Brief Title: Effect of the CFTR-modulating Triple Therapy Elexacaftor - Tezacaftor - Ivacaftor
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Alexander Schnell, Principle Investigator, University of Erlangen-Nürnberg Medical School
Other Study IDs: CF-Immuno
Record Dates: First submitted 2022-09-27; First posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Clinical parameters; Immune cell function
MeSH Terms: conditions — Cystic Fibrosis | interventions — elexacaftor, ivacaftor, tezacaftor drug combination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum Peripheral Mononuclear Blood Cells (PBMCs)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- longitudinal: Inclusion of patients with diagnosed CF prior ETI therapy, follow-up visit after 6 months
  Interventions: Drug: Elexacaftor / Ivacaftor / Tezacaftor
- under ETI: Patients with diagnosed CF already receiving ETI therapy for 6 months
  Interventions: Drug: Elexacaftor / Ivacaftor / Tezacaftor
- no ETI: Patients with diagnosed CF that have refused an ETI treatment or are not eligible for ETI therapy
- Healthy Individuals: Healthy, age- and gender-matched probands

INTERVENTIONS:
Drug: Elexacaftor / Ivacaftor / Tezacaftor — Elexacaftor / Ivacaftor / Tezacaftor is a triple drug therapy that modulates CFTR availability at (apical) cell membranes and increases opening probability.
  Other Names: ETI, Kaftrio®
  Groups: longitudinal; under ETI

SUMMARY:
The aim of this study is to investigate the frequency distribution, cytokine profile and function of peripheral, mononuclear leukocyte populations (monocytes, NK cells, T/B lymphocytes) and their correlation to clinical and biochemical parameters in patients with cystic fibrosis receiving CFTR modulatory triple therapy consisting of elexacaftor, tezacaftor and ivacaftor and to compare it with patients without CFTR modulatory therapy and healthy control subjects.

DETAILED DESCRIPTION:
The therapy of cystic fibrosis usually consists of an inhalative therapy with hy-pertonic saline and other mucolytics (e.g. dornase alpha) for secretolysis as well as a pancreatic enzyme replacement therapy. In recent years, however, the introduction of novel drugs, the so-called CFTR modulators, has revolutionized the previous treatment concept of a symptom-oriented therapy. Ivacaftor, which was approved by the FDA in 2012 for the treatment of patients with G551D mutation, causes a prolongation of the opening probability of the CFTR channel (CFTR potentiator) and was able to show a significant improvement in lung function in studies. By combining ivacaftor with the CFTR corrector lumacaftor, which improves the processing of the CFTR channel in the endoplasmic reticulum as well as its incorporation into the cell membrane, this therapeutic strategy has also been successfully tested for use in patients with F508del homozygous mutation. Also, the combination of ivacaftor with another CFTR corrector, tezacaftor, was approved for the treatment of patients with F508del heterozygous mutations in which the second mutation was classified as a mutation with residual activity and was able to show an increase in FEV1. The efficacy of this therapeutic approach was further enhanced by the combination of ivacaftor as a CFTR potentiator with tezacaftor and a next-generation CFTR corrector, elexacaftor; in the pivotal study, an improvement in FEV1 of an average of 14 points in untreated patients and 11 points in ivacaftor/tezacaftor-pretreated patients was demonstrated, as well as a significant decrease in hospitalizations due to pulmonary exacerbation. Since September 2020 in the European Union, this combination has been approved under the trade name Kaftrio® for the treatment of patients with F508del homozygous mutation or F508del heterozygous mutation and minimal function mutation. This form of therapy is based on a concept that comes closest to a causal therapy. In April 2021, the EMA granted approval for the drug for all patients older than 12 years and with evidence of at least one F508del mutation. In addition, the manufacturer applied for an extension of the approval in the EU for children aged 6-11 years based on the also very positive study results and received a positive decision from the European Medicines Agency (EMA) in November 2021. However, in addition to the clear role of the CFTR channel in epithelial tissues, it has been increasingly shown in recent years that the CFTR channel is also expressed by a variety of immune cells of the innate as well as the acquired immune system, such as neutrophils, macrophages, monocytes, and B and T lymphocytes. Its absence or dysfunction in cystic fibrosis seems to trigger a disturbed regulation or an exaggerated reaction of various immune responses.

ELIGIBILITY:
Inclusion Criteria:

* Patients (m/f/d) with molecularly genetically confirmed cystic fibrosis aged 6 years and older.
* Do not meet any of the exclusion criteria
* Written informed consent
* For study arm "Kaftrio® ongoing": Kaftrio® therapy for at least 6 months
* For study arm "Kaftrio® longitudinal": no Kaftrio® therapy started yet

Exclusion Criteria:

* Use of inhaled or systemic glucocorticoids as part of a permanent medication regimen
* Pregnancy

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients who are under the care of the CF Center Erlangen at the time of the study and who meet the inclusion criteria will be considered for the patient collective.
  Recruitment of healthy subjects will be performed during routine blood sampling in patients with pulmonary disease during outpatient appointments as well as during inpatient stays after prior informed consent has been obtained.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2020-12-30 (Actual); Primary Completion 2023-10-18 (Estimated); Study Completion 2023-10-18 (Estimated)

PRIMARY OUTCOMES:
Peripheral Blood Immunograms | prior ETI
  Relative and absolute peripheral blood immune cell count as determined by multicolor flow cytometry
Peripheral Blood Immunograms | 6 months ETI
  Relative and absolute peripheral blood immune cell count as determined by multicolor flow cytometry

SECONDARY OUTCOMES:
Shear Wave Velocity (SWV) | prior ETI
  Difference of mean/median SWV in treated vs. untreated patients as measured by Acoustic Radiation Force Impulse Imaging (ARFI)
Shear Wave Velocity (SWV) | 6 months ETI
  Difference of mean/median SWV in treated vs. untreated patients as measured by Acoustic Radiation Force Impulse Imaging (ARFI)
Attenuation Coefficient (AC) | prior ETI
  Difference of mean/median AC in treated vs. untreated pediatric patients (6-11 yrs) as measured by Ultrasound-guided attenuation parameter (UGAP)
Attenuation Coefficient (AC) | 6 months ETI
  Difference of mean/median AC in treated vs. untreated pediatric patients (6-11 yrs) as measured by Ultrasound-guided attenuation parameter (UGAP)
Serum bile acids | prior ETI
  Level of serum bile acids as measured by mass spectrometry
Serum bile acids | 6 months ETI
  Level of serum bile acids as measured by mass spectrometry
Respiratory function test (FEV1, FVC) | prior ETI
  Respiratory function test (FEV1, FVC) as measured by bodyplethysmography
Respiratory function test (FEV1, FVC) | 6 months ETI
  Respiratory function test (FEV1, FVC) as measured by bodyplethysmography
Blood cell count | prior ETI
  Blood cell count as defined in x10^3/µl
Blood cell count | 6 months ETI
  Blood cell count as defined in x10^3/µl
Erythrocytoid hemoglobin A1c | prior ETI
  Erythrocytoid hemoglobin A1c in %
Erythrocytoid hemoglobin A1c | 6 months ETI
  Erythrocytoid hemoglobin A1c in %
Plasma electrolytes | 6 months ETI
  Plasma electrolytes (Na, Cl) as defined by mmol/l
Liver transaminases | prior ETI
  Aspartate/Alanine aminotransferase (AST, ALt) as defined in U/l
Liver transaminases | 6 months ETI
  Aspartate/Alanine aminotransferase (AST, ALt) as defined in U/l
Plasmatic bilirubin | prior ETI
  Total and direct plasmatic bilirubin as defined in mg/dl
Plasmatic bilirubin | 6 months ETI
  Total and direct plasmatic bilirubin as defined in mg/dl
Prothrombin time | prior ETI
  Prothrombin time as defined by Quick percent
Prothrombin time | 6 months ETI
  Prothrombin time as defined by Quick percent
Coagulation factors | prior ETI
  Vitamin K- dependent coagulation factors (II, VII, IX, X) as measured in %
Coagulation factors | 6 months ETI
  Vitamin K- dependent coagulation factors (II, VII, IX, X) as measured in %
Plasmatic albumine | prior ETI
  Plasma levels of albumine (defined in g/dl)
Plasmatic albumine | 6 months ETI
  Plasma levels of albumine (defined in g/dl)
Plasmatic C-reactive proteine | prior ETI
  Plasmatic C-reactive proteine (defined in mg/l)
Plasmatic C-reactive proteine | 6 months ETI
  Plasmatic C-reactive proteine (defined in mg/l)
Plasmatic cholinesterase | prior ETI
  Plasmatic cholinesterase (defined in U/l)
Plasmatic cholinesterase | 6 months ETI
  Plasmatic cholinesterase (defined in U/l)
Plasmatic glutamate dehydrogenase | 6 months ETI
  Plasmatic glutamate dehydrogenase (defined in U/l)
Plasmatic creatinin | prior ETI
  Plasmatic creatinin (defined in mg/dl)
Plasmatic creatinin | 6 months ETI
  Plasmatic creatinin (defined in mg/dl)
Serum immunoglobulins | prior ETI
  Serum immunoglobulins G, A, M, E (defined in g/l)
Serum immunoglobulins | 6 months ETI
  Serum immunoglobulins G, A, M, E (defined in g/l)
Sweat chloride | prior ETI
  Sweat chloride level (defined in mmol/l)
Sweat chloride | 6 months ETI
  Sweat chloride level (defined in mmol/l)
BMI | prior ETI
  BMI in kg/m^2
BMI | 6 months ETI
  BMI in kg/m^2
Age | prior ETI
  Patients' age in years
Microbial colonization status | prior ETI
  Microbial colonization status as defined by microbiological reports
Microbial colonization status | 6 months ETI
  Microbial colonization status as defined by microbiological reports
Individual concomitant medication regime | prior ETI
  Individual concomitant medication regime
Individual concomitant medication regime | 6 months ETI
  Individual concomitant medication regime
Functional pulmonary magnetic resonance imaging | prior ETI
  Ventilation defect, perfusion defect, combined defects in longitudinal pediatric cohort (6-11 yrs)
Functional pulmonary magnetic resonance imaging | 6 months ETI
  Ventilation defect, perfusion defect, combined defects in longitudinal pediatric cohort (6-11 yrs)
Neutrophilic dihydrorhodamine assay | prior ETI
  Assay for determination of neutrophilic reactive oxygen species (measured as stimulation index)
Neutrophilic dihydrorhodamine assay | 6 months ETI
  Assay for determination of neutrophilic reactive oxygen species (measured as stimulation index)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Erlange, Department of Pediatrics, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keating D, Marigowda G, Burr L, Daines C, Mall MA, McKone EF, Ramsey BW, Rowe SM, Sass LA, Tullis E, McKee CM, Moskowitz SM, Robertson S, Savage J, Simard C, Van Goor F, Waltz D, Xuan F, Young T, Taylor-Cousar JL; VX16-445-001 Study Group. VX-445-Tezacaftor-Ivacaftor in Patients with Cystic Fibrosis and One or Two Phe508del Alleles. N Engl J Med. 2018 Oct 25;379(17):1612-1620. doi: 10.1056/NEJMoa1807120. Epub 2018 Oct 18. PMID 30334692
- [Background] Zemanick ET, Taylor-Cousar JL, Davies J, Gibson RL, Mall MA, McKone EF, McNally P, Ramsey BW, Rayment JH, Rowe SM, Tullis E, Ahluwalia N, Chu C, Ho T, Moskowitz SM, Noel S, Tian S, Waltz D, Weinstock TG, Xuan F, Wainwright CE, McColley SA. A Phase 3 Open-Label Study of Elexacaftor/Tezacaftor/Ivacaftor in Children 6 through 11 Years of Age with Cystic Fibrosis and at Least One F508del Allele. Am J Respir Crit Care Med. 2021 Jun 15;203(12):1522-1532. doi: 10.1164/rccm.202102-0509OC. PMID 33734030
- [Background] McDonald TV, Nghiem PT, Gardner P, Martens CL. Human lymphocytes transcribe the cystic fibrosis transmembrane conductance regulator gene and exhibit CF-defective cAMP-regulated chloride current. J Biol Chem. 1992 Feb 15;267(5):3242-8. PMID 1371114
- [Derived] Schnell A, Jungert J, Klett D, Hober H, Kaiser N, Ruppel R, Geppert A, Tremel C, Sobel J, Plattner E, Schmitt-Grohe S, Zirlik S, Strobel D, Neurath MF, Knieling F, Rauh M, Woelfle J, Hoerning A, Regensburger AP. Increase of liver stiffness and altered bile acid metabolism after triple CFTR modulator initiation in children and young adults with cystic fibrosis. Liver Int. 2023 Apr;43(4):878-887. doi: 10.1111/liv.15544. Epub 2023 Feb 28. PMID 36797990